CLINICAL TRIAL: NCT05222633
Title: Observation of Anti-vascular Endothelial Growth Factor Therapy in Exudative Age-related Macular Degeneration, Proliferative Diabetic Retinopathy, Macular Edema, and Choroidal Neovascularization.
Brief Title: Anti-VEGF in Real-world
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenbin Wei (Other)
Responsible Party: Sponsor-Investigator, Wenbin Wei, Director, Beijing Tongren Hospital
Organization: Beijing Tongren Hospital (Other)
Other Study IDs: Anti-VEGF in real-world
Record Dates: First submitted 2021-12-25; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Neovascular Age-related Macular Edema; Diabetic Macular Edema; Choroidal Neovascular Membrane; Non-proliferative Diabetic Retinopathy; Retinal Vein Occlusion; Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab; aflibercept; KH902 fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Neovascular age-related macular edema: Patients with new-onset and recurrent Neovascular age-related macular edema.
  Interventions: Drug: Ranibizumab; Drug: Aflibercept; Drug: Conbercept
- Diabetic macula edema: Patients with new-onset and recurrent diabetic macula edema
  Interventions: Drug: Ranibizumab; Drug: Aflibercept; Drug: Conbercept
- Non-proliferative diabetic retinopathy/proliferative diabetic retinopathy: Patients with new-onset and recurrent non-proliferative diabetic retinopathy/proliferative diabetic retinopathy
  Interventions: Drug: Ranibizumab; Drug: Aflibercept; Drug: Conbercept
- Retinal vein occlusions: Patients with new-onset and recurrent retinal vein occlusions
  Interventions: Drug: Ranibizumab
- Choroidal neovascularization: Patients with new-onset and recurrent choroidal neovascularization
  Interventions: Drug: Ranibizumab; Drug: Aflibercept; Drug: Conbercept

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5mg/0.05ml intravitreal injection
Drug: Aflibercept — Aflibercept 2.0mg/0.05ml intravitreal injection
  Groups: Choroidal neovascularization; Diabetic macula edema; Neovascular age-related macular edema; Non-proliferative diabetic retinopathy/proliferative diabetic retinopathy
Drug: Conbercept — Conbercept 0.5mg/0.05ml intravitreal injection
  Groups: Choroidal neovascularization; Diabetic macula edema; Neovascular age-related macular edema; Non-proliferative diabetic retinopathy/proliferative diabetic retinopathy

SUMMARY:
Anti-vascular endothelial growth factor therapy is the major intervention for treating ischemic retina diseases. According to FDA and China Food and Drug Administration, Ranibizumab, Aflibercept, and Conbercept are major types of anti-vascular endothelial growth factor therapy drugs. In the current study, the primary aim is to observe the visual acuity, anatomy effect of anti-vascular endothelial growth factor therapy in the real-world setting.

DETAILED DESCRIPTION:
Anti-vascular endothelial growth factor therapy is the major intervention for treating ischemic retina diseases, including neovascular age-related macular edema, diabetic macula edema/non-proliferative diabetic retinopathy / proliferative diabetic retinopathy, retinal vein occlusions related macular edema, and choroidal neovascularization secondary to multiple retinal diseases. According to FDA and China Food and Drug Administration, Ranibizumab, Aflibercept, and Conbercept are major types of anti-VEGF drugs. In the current study, the primary aim is to aim to observe the visual acuity, anatomy effect of anti-vascular endothelial growth factor therapy in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neovascular age-related macular edema (nAMD), diabetic macula edema (DME)/non-proliferative diabetic retinopathy (NPDR)/ proliferative diabetic retinopathy (PDR), retinal vein occlusions related macular edema, and choroidal neovascular (CNV) secondary to multiple retinal diseases.
* Undergo intravitreal anti-VEGF therapy

Exclusion Criteria:

* unable to receive OCT examination
* Severe corneal opacity, cataract that affect OCT examination

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular age-related macular edema (nAMD), diabetic macula edema (DME)/non-proliferative diabetic retinopathy (NPDR)/ proliferative diabetic retinopathy (PDR), retinal vein occlusions related macular edema, and choroidal neovascular (CNV) secondary to multiple retinal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  LogMAR visual acuity
Central subfield thickness | 1 year
  he central subfield is defined as the circular area 1 mm in diameter centered around the center point of the fovea

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, MD, Study Director — Beijing Tongren Hospital
Locations (1):
- Wen-Bin Wei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided